CLINICAL TRIAL: NCT02625207
Title: A Phase 1, Open-label, Parallel-group Study To Assess The Effect Of Cyp3a5 Genotype On The Pharmacokinetics Of Maraviroc And Cyp3a5-derived Metabolites With And Without Darunavir/Cobicistat In African-american And Caucasian Healthy Volunteers
Brief Title: THE EFFECT OF CYP3A5 GENOTYPE ON THE PHARMACOKINETICS OF MARAVIROC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4001110
Record Dates: First submitted 2015-10-20; First posted 2015-12-09 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Healthy Subjects
Keywords: Maraviroc, CYP3A5, pharmacokinetics, pharmacogenomics
MeSH Terms: interventions — Maraviroc; Darunavir; Cobicistat; cobicistat mixture with darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): African-Americans with No CYP3A5*1 alleles (poor metabolizer)
  Interventions: Drug: Maraviroc (Part 1); Drug: Maraviroc (Part 2); Drug: Darunavir/cobicistat (Part 2)
- Cohort 2 (Experimental): African-Americans with One CYP3A5*1 allele (intermediate metabolizer)
  Interventions: Drug: Maraviroc (Part 1)
- Cohort 3 (Experimental): African-Americans with Two CYP3A5*1 alleles (extensive metabolizer)
  Interventions: Drug: Maraviroc (Part 1); Drug: Maraviroc (Part 2); Drug: Darunavir/cobicistat (Part 2)
- Cohort 4 (Experimental): Caucasians with No CYP3A5*1 alleles (poor metabolizer)
  Interventions: Drug: Maraviroc (Part 1)

INTERVENTIONS:
Drug: Maraviroc (Part 1) — 300 mg twice daily x 5 days
  Other Names: Selzentry
Drug: Maraviroc (Part 2) — 150 mg once daily x 10 days
  Other Names: Selzentry
  Arms: Cohort 1; Cohort 3
Drug: Darunavir/cobicistat (Part 2) — 800/150 mg once daily x 10 days
  Other Names: Prezcobix
  Arms: Cohort 1; Cohort 3

SUMMARY:
This will be an open-label, parallel group, multiple dose study in approximately 48 healthy male or female subjects of African American and Caucasian self-reported race, to assess the effect of CYP3A5 genotype on the PK of MVC and CYP3A5-derived metabolites. Maraviroc and CYP3A5-derived metabolite PK will also be compared between African-Americans and Caucasians in subjects carrying two copies of the dysfunctional CYP3A5 alleles (*3, *6, and/or *7).

DETAILED DESCRIPTION:
This will be an open-label, parallel group, multiple dose study in approximately 48 healthy male or female subjects of African American and Caucasian self-reported race, to assess the effect of CYP3A5 genotype on the PK of MVC and CYP3A5-derived metabolites. Maraviroc and CYP3A5-derived metabolite PK will also be compared between African-Americans and Caucasians in subjects carrying two copies of the dysfunctional CYP3A5 alleles (*3, *6, and/or *7).

Dysfunctional genetic variants for CYP3A5, CYP3A4 and SLCO1B1 will be genotyped for subjects who participate in the pre-screening. Subjects who meet the inclusion/exclusion criteria for study participation will be placed into the study cohorts based on race and the number of functional (*1) and dysfunctional CYP3A5 alleles (*3, *6, and *7) CYP3A5 alleles.

Cohort 1 (n=12; African-American): No CYP3A5*1 alleles (poor metabolizer). Cohort 2 (n=12; African-American): One CYP3A5*1 allele (intermediate metabolizer).

Cohort 3 (n=12; African-American): Two CYP3A5*1 alleles (extensive metabolizer).

Cohort 4 (n=12; Caucasian): No CYP3A5*1 alleles (poor metabolizer).

Study Treatments:

Part 1 Days 1-5: Maraviroc 300 mg BID in fasted state (AM dose only on Day 5). Part 2 (Cohorts 1 and 3 only) Days 1-10: Maraviroc 150 mg QD plus darunavir/cobicistat 800/150 mg QD with food.

Pharmacokinetics of MVC, PF-6857639, PF-6857640 and other hydroxylated metabolites with formation mediated by CYP3A5 (if present) will be assessed on Part 1, Day 5 and Part 2, Days 10-11. Blood samples will be collected for a full PK profile.

Subjects will be confined to the Clinical Research Unit (CRU) the day prior to dosing on Day 1 (Day 0) and discharged on Part 1, Day 6 and on Part 2, Day 11 (Cohorts 1 and 3 only). Subjects enrolled into Cohorts 1 and 3 may be confined to the CRU without the need to be discharged between Part 1 and Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)
* Healthy female subjects and/or male subjects of African-American/Black or Caucasian race

Exclusion Criteria:

* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males
* Treatment with an investigational drug within 30 days
* Screening supine blood pressure <90 or >/=140 mm Hg (systolic) or <60 or >/= 90 mm Hg (diastolic), following at least 5 minutes of supine rest
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day
* Subjects who have a CYP3A4*22 allele and/or have a SLCO1B1 *5 or *15 allele

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-03-26 (Actual); Study Completion 2016-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Vourvahis M, McFadyen L, Nepal S, Valluri SR, Fang A, Fate GD, Wood LS, Marshall JC, Chan PLS, Nedderman A, Haynes J, Savage ME, Clark A, Smith KY, Heera J. No Clinical Impact of CYP3A5 Gene Polymorphisms on the Pharmacokinetics and/or Efficacy of Maraviroc in Healthy Volunteers and HIV-1-Infected Subjects. J Clin Pharmacol. 2019 Jan;59(1):139-152. doi: 10.1002/jcph.1306. Epub 2018 Sep 7. PMID 30192390
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001110&StudyName=A%20Phase%201%2C%20Open-label%2C%20Parallel-group%20Study%20To%20Assess%20The%20Effect%20Of%20Cyp3a5%20Genotype%20On%20The%20Pharmacokinetics%20Of%20Maraviroc%20And%20Cyp3a5-derived%20Metabolites%20With%20And%20Without%20Darunavir%2Fcobicistat%20In%20African-american%20And%20Caucasian%20Healthy%20Volunteers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in two parts (Part 1 and 2). Participants were assigned to treatment into 4 cohorts in Part 1 (Cohort 1, 2, 3, 4) and into 2 cohorts in part 2 (Cohort 1, 3).
Groups:
- Part 1 and Part 2: Cohort 1 -No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 300 milligram (mg) tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1, followed by maraviroc 150 mg tablet once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2.
- Part 1: Cohort 2 - One CYP3A5*1 Allele: African-American participants with one CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
- Part 1 and 2: Cohort 3 - Two CYP3A5*1 Alleles: African-American participants with two CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1, followed by maraviroc 150 mg tablet once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2.
- Part 1: Cohort 4 - No CYP3A5*1 Alleles: Caucasian participants with no CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
Period: Part 1 (6 Days)
Arm/Group | Part 1 and Part 2: Cohort 1 -No CYP3A5*1 Alleles | Part 1: Cohort 2 - One CYP3A5*1 Allele | Part 1 and 2: Cohort 3 - Two CYP3A5*1 Alleles | Part 1: Cohort 4 - No CYP3A5*1 Alleles
Started | 11 | 12 | 12 | 12
Completed | 11 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 (11 Days)
Arm/Group | Part 1 and Part 2: Cohort 1 -No CYP3A5*1 Alleles | Part 1: Cohort 2 - One CYP3A5*1 Allele | Part 1 and 2: Cohort 3 - Two CYP3A5*1 Alleles | Part 1: Cohort 4 - No CYP3A5*1 Alleles
Started | 11 | 0 (Part 2 was conducted only in Cohorts 1 and 3, as pre-specified in protocol.) | 12 | 0 (Part 2 was conducted only in Cohorts 1 and 3, as pre-specified in protocol.)
Completed | 11 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Part 1 and Part 2: Cohort 1 -No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1, followed by maraviroc 150 mg tablet once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2.
- Total: Total of all reporting groups
Arm/Group | Part 1 and Part 2: Cohort 1 -No CYP3A5*1 Alleles | Part 1: Cohort 2 - One CYP3A5*1 Allele | Part 1 and 2: Cohort 3 - Two CYP3A5*1 Alleles | Part 1: Cohort 4 - No CYP3A5*1 Alleles | Total
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (9.7) | 38.3 (10.4) | 34.6 (11.4) | 48.2 (6) | 39.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 4
  Male | 9 | 12 | 11 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under The Plasma Concentration-Time Curve From Time 0 to 12 Hours (AUC [0-12]) of Maraviroc
Description: AUC (0-12) is the area under the plasma concentration versus time curve from time zero (pre-dose) to 12 hours post-dose.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: Pharmacokinetic (PK) parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Cohort 1- No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
- Cohort 2- One CYP3A5*1 Allele: African-American participants with one CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
- Cohort 3- Two CYP3A5*1 Alleles: African-American participants with two CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
- Cohort 4- No CYP3A5*1 Alleles: Caucasian participants with no CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 3441 (24) | 2954 (23) | 2181 (27) | 2947 (23)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.1318, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 116.73, 90% CI 2-sided [98.55 to 138.26]
Statistical Analysis 2: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Test type: Superiority or Other; p = 0.1369, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 85.85, 90% CI 2-sided [72.48 to 101.68]
Statistical Analysis 3: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 63.38, 90% CI 2-sided [53.51 to 75.07]
Statistical Analysis 4: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 73.83, 90% CI 2-sided [62.57 to 87.13]
Statistical Analysis 5: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis; Adjusted Geometric Mean ratio = 73.99, 90% CI 2-sided [62.70 to 87.31]

2. Primary Outcome: Part 2: Area Under The Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC [0-24]) of Maraviroc
Description: AUC (0-24) is the area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post-dose.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose on Day 10
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of primary interest. Data for Part 2 was planned to be analyzed only in Cohorts 1 and 3, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Cohort 1- No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 150 mg tablet orally once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2 .
- Cohort 3- Two CYP3A5*1 Alleles: African-American participants with two CYP3A5*1 alleles, received maraviroc 150 mg tablet orally once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2.
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
ng*hr/mL | 4413 (20) | 3645 (25)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0531, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 82.59, 90% CI 2-sided [70.33 to 96.98]

3. Primary Outcome: Part 1: Metabolite to Parent Ratio for Area Under the Concentration-Time Curve From Time 0 to 12 Hours for Maraviroc and Its Metabolites (MRAUC12)
Description: MRAUC12 is the ratio of AUC12 of maraviroc to AUC12 of maraviroc's metabolites. Metabolites of Maraviroc included PF-6857639, PF-6857640, PF-06927572 and PF-06927573. AUC12 is the area under the plasma concentration-time profile from time 0 to 12 hours post-dose.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: PK parameter analysis set included all randomized and treated participants who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ratio
  PF-6857639 | 0.02172 (31) | 0.03564 (27) | 0.04312 (32) | 0.01585 (24)
  PF-6857640 | 0.02577 (11) | 0.02621 (27) | 0.02797 (32) | 0.02338 (14)
  PF-06927572 | 0.02766 (19) | 0.02908 (35) | 0.02795 (37) | 0.02774 (29)
  PF-06927573 | 0.02048 (14) | 0.02427 (38) | 0.02040 (27) | 0.02099 (21)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -6857639 was estimated and reported; Test type: Superiority or Other; p = 0.0106, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 137.07, 90% CI 2-sided [112.40 to 167.15]
Statistical Analysis 2: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Statistical analysis of PF -6857639 was estimated and reported; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 164.06, 90% CI 2-sided [134.54 to 200.06]
Statistical Analysis 3: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -6857639 was estimated and reported; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 198.49, 90% CI 2-sided [162.77 to 242.05]
Statistical Analysis 4: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -6857639 was estimated and reported; Test type: Superiority or Other; p = 0.1061, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 120.99, 90% CI 2-sided [99.65 to 146.90]
Statistical Analysis 5: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -6857639 was estimated and reported; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 272.07, 90% CI 2-sided [224.08 to 330.33]
Statistical Analysis 6: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -6857640 was estimated and reported; Test type: Superiority or Other; p = 0.3081, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 110.22, 90% CI 2-sided [94.05 to 129.18]
Statistical Analysis 7: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Statistical analysis of PF -6857640 was estimated and reported; Test type: Superiority or Other; p = 0.8583, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 101.71, 90% CI 2-sided [86.79 to 119.20]
Statistical Analysis 8: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -6857640 was estimated and reported; Test type: Superiority or Other; p = 0.3913, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 108.52, 90% CI 2-sided [92.60 to 127.17]
Statistical Analysis 9: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -6857640 was estimated and reported; Test type: Superiority or Other; p = 0.4866, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 106.69, 90% CI 2-sided [91.36 to 124.60]
Statistical Analysis 10: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -6857640 was estimated and reported; Test type: Superiority or Other; p = 0.0590, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 119.61, 90% CI 2-sided [102.42 to 139.69]
Statistical Analysis 11: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -06927572 was estimated and reported; Test type: Superiority or Other; p = 0.9816, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 99.70, 90% CI 2-sided [80.47 to 123.53]
Statistical Analysis 12: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Statistical analysis of PF -06927572 was estimated and reported; Test type: Superiority or Other; p = 0.6974, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 105.12, 90% CI 2-sided [84.84 to 130.24]
Statistical Analysis 13: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -06927572 was estimated and reported; Test type: Superiority or Other; p = 0.9363, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 101.03, 90% CI 2-sided [81.54 to 125.18]
Statistical Analysis 14: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -06927572 was estimated and reported; Test type: Superiority or Other; p = 0.7520, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 96.11, 90% CI 2-sided [77.94 to 118.52]
Statistical Analysis 15: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -06927572 was estimated and reported; Test type: Superiority or Other; p = 0.9536, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 100.73, 90% CI 2-sided [81.69 to 124.22]
Statistical Analysis 16: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -06927573 was estimated and reported; Test type: Superiority or Other; p = 0.8241, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 97.60, 90% CI 2-sided [81.28 to 117.18]
Statistical Analysis 17: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Statistical analysis of PF -06927573 was estimated and reported; Test type: Superiority or Other; p = 0.1261, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 118.50, 90% CI 2-sided [98.69 to 142.28]
Statistical Analysis 18: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -06927573 was estimated and reported; Test type: Superiority or Other; p = 0.9708, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 99.60, 90% CI 2-sided [82.95 to 119.59]
Statistical Analysis 19: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Statistical analysis of PF -06927573 was estimated and reported; Test type: Superiority or Other; p = 0.1099, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 84.05, 90% CI 2-sided [70.29 to 100.52]
Statistical Analysis 20: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Statistical analysis of PF -06927573 was estimated and reported; Test type: Superiority or Other; p = 0.7913, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 97.21, 90% CI 2-sided [81.29 to 116.25]

4. Secondary Outcome: Part 1: Average Plasma Concentration (Cavg) of Maraviroc
Description: Cavg is the average plasma concentration of maraviroc during the 0 to 12 hour time period. It was calculated as area under the plasma concentration-time curve from 0 to 12 hours (AUC [0-12]) divided by 12.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
nanogram per milliliter (ng/mL) | 286.8 (24) | 246.2 (23) | 181.6 (27) | 245.8 (23)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.1338, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 116.65, 90% CI 2-sided [98.47 to 138.18]
Statistical Analysis 2: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Test type: Superiority or Other; p = 0.1370, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 85.84, 90% CI 2-sided [72.46 to 101.68]
Statistical Analysis 3: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 63.34, 90% CI 2-sided [53.47 to 75.04]
Statistical Analysis 4: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis; Adjusted Geometric Mean ratio = 73.79, 90% CI 2-sided [62.53 to 87.09]
Statistical Analysis 5: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0037, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 73.89, 90% CI 2-sided [62.61 to 87.20]

5. Secondary Outcome: Part 2: Average Plasma Concentration (Cavg) of Maraviroc
Description: Cavg is the average plasma concentration of maraviroc during the 0 to 24 hour time period. It was calculated as area under the plasma concentration-time curve from 0 to 24 hours (AUC [0-24]) divided by 24.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose on Day 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1- No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 150 mg tablet orally once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2.
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
ng/mL | 184.1 (20) | 151.7 (25)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0507, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 82.42, 90% CI 2-sided [70.20 to 96.77]

6. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Maraviroc
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng/mL | 863.9 (29) | 754.0 (29) | 529.0 (34) | 731.0 (33)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.1997, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 118.19, 90% CI 2-sided [95.26 to 146.63]
Statistical Analysis 2: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Test type: Superiority or Other; p = 0.2947, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 87.28, 90% CI 2-sided [70.34 to 108.28]
Statistical Analysis 3: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 61.23, 90% CI 2-sided [49.35 to 75.97]
Statistical Analysis 4: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 70.16, 90% CI 2-sided [56.81 to 86.63]
Statistical Analysis 5: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0135, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 72.37, 90% CI 2-sided [58.60 to 89.36]

7. Secondary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Maraviroc
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose on Day 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 3- Two CYP3A5*1 Alleles: African-American participants with two CYP3A5*1 alleles, received maraviroc 150 mg tablet orally once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2 .
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
ng/mL | 633.6 (37) | 432.9 (53)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0505, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 68.32, 90% CI 2-sided [49.81 to 93.71]

8. Secondary Outcome: Part 1: Plasma Concentration of Maraviroc at 12 Hours Post-dose
Time Frame: 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng/mL | 59.84 (36) | 63.09 (27) | 45.32 (35) | 63.10 (24)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.6761, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 94.83, 90% CI 2-sided [76.70 to 117.24]
Statistical Analysis 2: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 2- One CYP3A5*1 Allele; Test type: Superiority or Other; p = 0.6771, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 105.43, 90% CI [85.28 to 130.35]
Statistical Analysis 3: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0331, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 75.74, 90% CI 2-sided [61.26 to 93.64]
Statistical Analysis 4: Comparison: Cohort 2- One CYP3A5*1 Allele vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0104, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 71.84, 90% CI 2-sided [58.38 to 88.40]
Statistical Analysis 5: Comparison: Cohort 3- Two CYP3A5*1 Alleles vs Cohort 4- No CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.0104, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 71.82, 90% CI 2-sided [58.37 to 88.39]

9. Secondary Outcome: Part 2: Plasma Concentration of Maraviroc at 24 Hours Post-dose
Time Frame: 24 hours post-dose on Day 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
ng/mL | 56.56 (20) | 56.34 (30)
Statistical Analysis 1: Comparison: Cohort 1- No CYP3A5*1 Alleles vs Cohort 3- Two CYP3A5*1 Alleles; Test type: Superiority or Other; p = 0.9713, Mixed Models Analysis; Adjusted Geometric Mean Ratio = 99.62, 90% CI 2-sided [83.07 to 119.45]

10. Secondary Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Maraviroc
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
hour | 3.00 [2.00 to 4.00] | 2.00 [0.500 to 3.00] | 2.00 [0.517 to 4.00] | 2.01 [0.500 to 3.05]

11. Secondary Outcome: Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Maraviroc
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24 hours post-dose on Day 10
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
hour | 3.00 [1.07 to 6.00] | 3.02 [1.00 to 6.02]

12. Secondary Outcome: Part 1: Area Under The Plasma Concentration-Time Curve From Time 0 to 12 Hours (AUC [0-12]) of Metabolites of Maraviroc
Description: AUC (0-12) is the area under the plasma concentration versus time curve from time zero (pre-dose) to 12 hours post-dose. Metabolites of maraviroc included PF-6857639, PF-6857640, PF-06927572 and PF-06927573.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng*hr/mL
  PF-6857639 | 77.09 (32) | 108.7 (44) | 96.98 (29) | 48.24 (32)
  PF-6857640 | 91.42 (22) | 79.92 (44) | 62.86 (26) | 71.15 (23)
  PF-06927572 | 98.14 (23) | 88.63 (49) | 62.80 (28) | 84.32 (33)
  PF-06927573 | 72.67 (28) | 73.92 (53) | 45.86 (27) | 63.88 (28)

13. Secondary Outcome: Part 1: Average Plasma Concentration (Cav) of Metabolites of Maraviroc
Description: Cavg is the average plasma concentration of metabolites of maraviroc during the 0 to 12 hour time period. It was calculated as area under the plasma concentration-time curve from 0 to 12 hours (AUC [0-12]) divided by 12. Metabolites of maraviroc included PF-6857639, PF-6857640, PF-06927572 and PF-06927573.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng/mL
  PF-6857639 | 6.420 (32) | 9.049 (44) | 8.074 (29) | 4.018 (32)
  PF-6857640 | 7.615 (22) | 6.658 (44) | 5.239 (26) | 5.930 (23)
  PF-06927572 | 8.179 (23) | 7.383 (49) | 5.232 (28) | 7.029 (33)
  PF-06927573 | 6.056 (28) | 6.165 (53) | 3.821 (27) | 5.323 (28)

14. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Metabolites of Maraviroc
Description: Metabolites of maraviroc included PF-6857639, PF-6857640, PF-06927572 and PF-06927573.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng/mL
  PF-6857639 | 18.14 (23) | 24.18 (55) | 20.52 (34) | 11.22 (37)
  PF-6857640 | 21.95 (28) | 18.96 (56) | 15.00 (30) | 16.48 (28)
  PF-06927572 | 22.88 (18) | 20.67 (58) | 15.31 (32) | 19.91 (35)
  PF-06927573 | 17.39 (32) | 17.64 (66) | 10.86 (34) | 15.27 (35)

15. Secondary Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Metabolites of Maraviroc
Description: Metabolites of maraviroc included PF-6857639, PF-6857640, PF-06927572 and PF-06927573.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 9, 12 hours post-dose on Day 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
hour
  PF-6857639 | 3.00 [1.00 to 4.00] | 2.00 [0.500 to 3.00] | 2.00 [0.533 to 4.00] | 3.00 [0.500 to 4.00]
  PF-6857640 | 3.00 [1.00 to 4.00] | 2.00 [0.500 to 3.02] | 2.00 [0.533 to 4.00] | 3.00 [1.00 to 4.00]
  PF-06927572 | 3.00 [1.00 to 4.00] | 2.00 [0.500 to 3.00] | 1.52 [0.500 to 4.00] | 3.00 [1.00 to 4.00]
  PF-06927573 | 3.00 [1.00 to 4.00] | 2.00 [0.500 to 3.00] | 2.00 [0.567 to 4.00] | 3.00 [1.00 to 4.00]

16. Secondary Outcome: Part 1: Plasma Concentration of Metabolites of Maraviroc at 12 Hour Post-dose
Description: Metabolites of maraviroc included PF-6857639, PF-6857640, PF-06927572 and PF-06927573.
Time Frame: 12 hour post-dose on Day 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng/mL
  PF-6857639 | 0.6249 (7399) | 2.748 (43) | 2.226 (32) | 0.9213 (38)
  PF-6857640 | 0.6290 (7164) | 1.658 (40) | 1.134 (29) | 1.300 (33)
  PF-06927572 | 0.6242 (7051) | 1.752 (45) | 1.071 (29) | 1.385 (40)
  PF-06927573 | 0.5396 (6283) | 1.629 (55) | 0.8550 (26) | 1.175 (32)

17. Secondary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 6 days that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to end of study (up to 6 days)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
participants
  AEs | 3 | 0 | 0 | 3
  SAEs | 0 | 0 | 0 | 0

18. Secondary Outcome: Part 2: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 11 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to end of study (up to 11 days)
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Data for Part 2 was planned to be analyzed only in Cohorts 1 and 3, as pre specified in protocol.
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
participants
  AEs | 2 | 1
  SAEs | 0 | 0

19. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for clinically significant vital sign abnormalities included supine/sitting pulse rate of less than (<) 40 beats per minute (bpm) or greater than (>)120 bpm, standing pulse rate of <40 bpm or >140 bpm, supine systolic blood pressure (SBP) and standing SBP of <90 millimeter of mercury (mm Hg), greater than or equal to (>=) 30 mm Hg, supine diastolic blood pressure (DBP) and standing DBP of <50 mm Hg, >=20 mm Hg.
Time Frame: Baseline up to Day 6
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for clinically significant vital sign abnormalities included supine/sitting pulse rate of <40 bpm or >120 bpm, standing pulse rate of <40 bpm or >140 bpm, supine SBP and standing SBP of <90 mm Hg, >=30 mm Hg, supine DBP and standing DBP of <50 mm Hg, >=20 mm Hg.
Time Frame: Baseline up to Day 11
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
participants | 0 | 0

21. Secondary Outcome: Part 1: Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: Maximum PR interval of >=300 milliseconds (msec), maximum QRS interval >=140 msec, maximum QTCF interval (Fridericia's correction) of 450 to <480 msec, 480 to <500 msec and >=500 msec, maximum increase of >=25 percent for baseline values of >200 msec and >=50 percent for baseline values of less than or equal to (<=) 200 msec for PR interval, maximum increase from baseline of >=50 percent for QRS interval, maximum increase from baseline of >=30 msec to <60 msec and maximum increase from baseline of >60 msec in QTCF interval (Fridericia's Correction).
Time Frame: Baseline up to Day 6
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Part 2: Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: Maximum PR interval of >=300 msec, maximum QRS interval >=140 msec, maximum QTCF interval (Fridericia's correction) of 450 to <480 msec, 480 to <500 msec and >=500 msec, maximum increase of >=25 percent for baseline values of >200 msec and >=50 percent for baseline values of <=200 msec for PR interval, maximum increase from baseline of >=50 percent for QRS interval, maximum increase from baseline of >=30 msec to <60 msec and maximum increase from baseline of >60 msec in QTCF interval (Fridericia's Correction).
Time Frame: Baseline up to Day 11
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
participants | 0 | 0

23. Secondary Outcome: Part 1: Number of Participants With Laboratory Abnormalities
Description: Criteria: Hemoglobin; hematocrit; red blood cell count: <0.8*lower limit of normal, (LLN), mean corpuscular volume; mean corpuscular hemoglobin concentration; mean platelet volume:<0.9*LLN or >1.1* upper limit of normal (ULN), platelet: <0.5*LLN or >1.75*ULN, white blood cells <0.6*LLN or >1.5*ULN, lymphocyte; neutrophil: <0.8*LLN or >1.2*ULN, basophil; eosinophil; monocyte:>1.2*ULN, bilirubin (total, direct, indirect) >1.5*ULN, aspartate aminotransferase; alanine aminotransferase; alkaline phosphatase:>3.0*ULN, total protein; albumin:<0.8*LLN or >1.2*ULN; creatinine: >1.3*ULN, uric acid>1.2*ULN, sodium<0.95*LLN or >1.05*ULN, potassium; chloride; calcium; bicarbonate:<0.9*LLN or >1.1*ULN, glucose <0.6*LLN or >1.5*ULN, urine specific gravity <1.003, urine pH <4.5 or >8, urine glucose or ketones (qualitative) >=1, urine protein; urine blood/hemoglobin >=1, urobilinogen; bilirubin; nitrite; leukocyte esterase >=1.
Time Frame: Baseline up to Day 6
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 2- One CYP3A5*1 Allele | Cohort 3- Two CYP3A5*1 Alleles | Cohort 4- No CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12 | 12 | 12
participants | 1 | 5 | 0 | 2

24. Secondary Outcome: Part 2: Number of Participants With Laboratory Abnormalities
Description: Criteria: Hemoglobin; hematocrit; red blood cell count: <0.8*LLN, mean corpuscular volume; mean corpuscular hemoglobin concentration; mean platelet volume: <0.9*LLN or >1.1*ULN, platelet: <0.5*LLN or >1.75*ULN, white blood cells <0.6*LLN or >1.5*ULN, lymphocyte; neutrophil: <0.8*LLN or >1.2*ULN, basophil; eosinophil; monocyte: >1.2*ULN, bilirubin (total, direct, indirect) >1.5*ULN, aspartate aminotransferase; alanine aminotransferase; alkaline phosphatase: >3.0*ULN, total protein; albumin: <0.8*LLN or >1.2*ULN; creatinine: >1.3*ULN, uric acid >1.2*ULN, sodium<0.95*LLN or >1.05*ULN, potassium; chloride; calcium; bicarbonate:<0.9*LLN or >1.1*ULN, glucose <0.6*LLN or >1.5*ULN, urine specific gravity <1.003, urine pH <4.5 or >8, urine glucose or ketones (qualitative) >=1, urine protein; urine blood/hemoglobin >=1, urobilinogen; bilirubin; nitrite; leukocyte esterase >=1.
Time Frame: Baseline up to Day 11
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Cohort 1- No CYP3A5*1 Alleles | Cohort 3- Two CYP3A5*1 Alleles
Number analyzed (Participants) | 11 | 12
participants | 1 | 3

ADVERSE EVENTS:
Description: Adverse events were collected and reported for Part 1 and Part 2 separately.
Groups:
- Part 1: Cohort 1- No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
- Part 1: Cohort 2- One CYP3A5*1 Allele; Part 1: Cohort 3- Two CYP3A5*1 Alleles: African-American participants with two CYP3A5*1 alleles, received maraviroc 300 mg tablet orally twice daily from Day 1 to Day 4 and once only in the morning of Day 5 in Part 1.
- Part 2: Cohort 1- No CYP3A5*1 Alleles: African-American participants with no CYP3A5*1 alleles, received maraviroc 150 mg tablet orally once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2 .
- Part 2: Cohort 3- Two CYP3A5*1 Alleles: African-American participants with two CYP3A5*1 alleles, received maraviroc 150 mg tablet orally once daily along with darunavir/cobicistat 800/150 mg tablet once daily from Day 1 to Day 10 in Part 2 .
Arm/Group | Part 1: Cohort 1- No CYP3A5*1 Alleles | Part 1: Cohort 2- One CYP3A5*1 Allele | Part 1: Cohort 3- Two CYP3A5*1 Alleles | Part 1: Cohort 4 - No CYP3A5*1 Alleles | Part 2: Cohort 1- No CYP3A5*1 Alleles | Part 2: Cohort 3- Two CYP3A5*1 Alleles
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 3/11 | 0/12 | 0/12 | 3/12 | 2/11 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort 1- No CYP3A5*1 Alleles (N=11) | Part 1: Cohort 2- One CYP3A5*1 Allele (N=12) | Part 1: Cohort 3- Two CYP3A5*1 Alleles (N=12) | Part 1: Cohort 4 - No CYP3A5*1 Alleles (N=12) | Part 2: Cohort 1- No CYP3A5*1 Alleles (N=11) | Part 2: Cohort 3- Two CYP3A5*1 Alleles (N=12)
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
As per change in planned analysis, calculation of metabolite PK parameters and statistical analyses were not conducted in Part 2, since substantial number of PK samples were below limit of quantitation, considered as non-reliable by investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.